CLINICAL TRIAL: NCT04911621
Title: Adjuvant Dendritic Cell Immunotherapy Complementing Conventional Therapy for Pediatric Patients With High-grade Glioma and Diffuse Intrinsic Pontine Glioma
Brief Title: Adjuvant Dendritic Cell Immunotherapy for Pediatric Patients With High-grade Glioma or Diffuse Intrinsic Pontine Glioma
Acronym: ADDICT-pedGLIO
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Kom Op Tegen Kanker (Other); Stichting Semmy (Unknown); Olivia Hendrickx research Fund vzw (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCRG19-002
Record Dates: First submitted 2021-04-30; First posted 2021-06-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: High Grade Glioma; Diffuse Intrinsic Pontine Glioma
Keywords: childhood glioma; dendritic cells; adjuvant therapy; immunotherapy; Wilms' tumor protein 1
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Intervention Model Description: Both newly diagnosed patients and patients who previously underwent anti-glioma treatment are eligible for the study, provided they comply with all in- and exclusion criteria. The study hence consists of two strata, newly diagnosed patients are included in stratum A, while pre-treated patients are included in stratum B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratum A (newly diagnosed) (Experimental): Dendritic cell vaccination plus temozolomide-based chemoradiotherapy
  Interventions: Biological: Dendritic cell vaccination + temozolomide-based chemoradiation
- Stratum B (prior treatment) (Experimental): Dendritic cell vaccination plus optional conventional anti-glioma treatment (in line with standard-of-care practice, at the investigator's discretion)
  Interventions: Biological: Dendritic cell vaccination +- conventional next-line treatment

INTERVENTIONS:
Biological: Dendritic cell vaccination + temozolomide-based chemoradiation — 1. Leukocyte apheresis (before chemoradiation): for dendritic cell (DC) vaccine production.
  2. Chemoradiation (1st part standard treatment, initiated as soon as the patient's hematological blood values are adequate after apheresis, but no later than 6 weeks after surgery or confirmed diagnosis): 1.8 Gy once daily 5 days/week for 6 weeks with 90 mg/m² temozolomide daily from the first until the last day of radiotherapy.
  3. Induction immunotherapy: intradermal vaccination with autologous Wilms' tumor-1 (WT1) mRNA-loaded DCs weekly (-1 day, +2 days) for 3 weeks, starting ≥ 1 week after radiotherapy.
  4. Chemo-immunotherapy: 150-200 mg/m²/d temozolomide days 1-5 every 28 days +/- 3 days (max. 6 months, 2nd part standart treatment) starting ≥3 days after the third vaccine of the induction immunotherapy + DC vaccination on day 21±3 days of every 28-day cycle.
  Arms: Stratum A (newly diagnosed)
Biological: Dendritic cell vaccination +- conventional next-line treatment — 1. Leukocyte apheresis (upon recovery of hematological blood values following previous anti-glioma treatments and ≥ 4 weeks after the last dose of any investigational agent): for DC vaccine production.
  2. Induction immunotherapy: intradermal vaccination with autologous WT1 mRNA-loaded DCs weekly (-1 day, +2 days) for 3 weeks, starting ≥ 4 weeks after apheresis.
  3. Booster immunotherapy: 6 DC booster vaccinations administered at regular intervals (+- 4 weeks), starting ≥ 3 weeks after the last induction vaccine.
  4. (Optional) Concomitant conventional anti-glioma treatment: The decision to continue or re-initiate conventional anti-glioma treatment, and, if applicable, its dose and scheme, are at the Investigator's discretion and will depend on the patient's previous treatment scheme and condition.
  Arms: Stratum B (prior treatment)

SUMMARY:
Childhood aggressive gliomas are rare brain tumors with very poor prognosis. Due to the tumor's location and infiltrative nature, surgical removal is not always possible, and even when resection is performed and combined with chemo- and/or radiotherapy, tumor cells frequently persist, eventually giving rise to tumor recurrence. A promising strategy to eradicate persisting tumor cells is vaccination with dendritic cells (DC). DC are immune cells that play an important role in organizing the body's defense against cancer. The goal of DC vaccination is to activate these natural anti-tumor defense mechanisms to delay or prevent tumor progression or recurrence. Previous clinical studies have demonstrated that DC vaccination is well-tolerated, safe and capable of eliciting tumorspecific immunity.

A clinical study including 10 pediatric patients (aged ≥ 12 months and < 18 years at the time of signing the informed consent) with brain (stem) tumors is initiated at the Antwerp University Hospital to investigate intradermal vaccination with WT1 mRNA-loaded autologous monocyte-derived DCs, either combined with first-line chemoradiation treatment or administered as adjuvant therapy following previous therapies. The general objective of this phase I/II clinical study is (1) to demonstrate that WT1-targeted DC vaccine production and administration in pediatric patients with HGG and DIPG, either combined with first-line chemoradiation treatment or administered as adjuvant therapy following previous therapies, is feasible and safe, (2) to study vaccine-induced immune responses, (3) to document patients' quality of life and clinical outcome for comparison with current patients' outcome allowing indication of the added value.

DETAILED DESCRIPTION:
1. Overview of the study treatment scheme

   1.1 Newly diagnosed HGG and DIPG patients (stratum A)

   Patients will be screened and registered in the study following diagnosis, which is based on either histological confirmation or radiographic criteria. Maximal safe resection prior to study entry is strongly recommended, but not required.

   Eligible patients will undergo leukapheresis prior to temozolomide-based chemoradiation and subsequent chemo-immunotherapy with maintenance temozolomide and autologous WT1 mRNA-loaded DC vaccination. Chemoradiation with subsequent maintenance temozolomide is considered best available treatment and therefore not considered investigational. The investigational treatment, i.e. adjuvant DC vaccination, is administered in 2 phases:
   * an induction phase, consisting of 3 weekly (-1 day, +2 days) DC vaccines, which is initiated after chemoradiation, but before maintenance temozolomide therapy, and
   * a booster phase, consisting of 6 4-weekly (±3 days) DC vaccines, which are administered during temozolomide maintenance cycles.

   1.2 Non-treatment naïve HGG and DIPG patients (stratum B)

   Patients who have undergone previous anti-glioma treatments can be included in the study, provided they are eligible according to the in- and exclusion criteria.

   The decision to start, continue or re-initiate conventional anti-glioma treatment, including radio- and/or chemotherapy, and, if applicable, the treatment dose and scheme, are at the Investigator's discretion. The backbone DC immunotherapy scheme for the induction and booster phase will be maintained with minor modifications:
   * during the induction phase, 3 DC vaccines will be administered on a weekly (-1 day, +2 days) basis
   * during the booster phase, 6 DC vaccines will be administered at regular intervals. It is recommended that the time between subsequent vaccinations is no longer than 4 weeks

   1.3 Continuation of DC vaccination

   While the study treatment schedule consists of 9 DC vaccinations (i.e. 3 induction and 6 booster vaccines), continuation of DC vaccination after the booster phase is allowed, on the conditions that (1) the Investigator judges that the participant's clinical situation justifies additional vaccinations, (2) consent for continuation of DC vaccination of the parents/guardian and the participant (if aged 12 years or older) has been obtained, and (3) residual vaccine aliquots are available.
2. Response assessment

   Disease evolution will be assessed radiologically according to the Response Assessment in Neuro-Oncology (RANO) criteria. In addition, blood samples will be collected for immunomonitoring purposes on the day of the first, fourth and seventh DC vaccine. Tumor resection or biopsy specimens, if available, will be used for local immunological and biomarker analysis. At regular time points throughout the study scheme, parents and participants will be asked to fill out questionnaires on general and disease-specific quality-of-life, as well as on executive function.
3. Follow-up

Patients will be followed-up until 90 days after administration of the final DC vaccine or 24 months after study entry, whichever occurs later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of

  * High grade glioma (WHO grade III or IV), histologically verified
  * Diffuse Intrinsic Pontine Glioma, verified by radiologic criteria (magnetic resonance imaging (MRI)) or by histology. A biopsy is not required but recommended.
* Aged ≥ 12 months and < 18 years at the time of signing the informed consent
* Body weight ≥ 10 kg
* Lansky score (for patients < 16 years) or Karnofsky score (for patients ≥ 16 years) of ≥ 50
* Reasonable life expectancy ≥ 8 weeks, as estimated by the treating physician
* Adequate hematological blood values and sufficient recovery from treatment-related toxicities (> grade 1) following previous anti-glioma treatments, as judged by the treating physician
* Written informed consent of parents or legal guardian. Written informed consent of patients aged 12 years or older (written informed consent of patients younger than 12 years is optional).
* Willing and able to comply with the protocol, as judged by the treating physician
* Female patients of child bearing potential must have a negative serum or urine pregnancy test at the time of screening. Female patients of child bearing potential and male patients must agree to use effective contraception before, during and for at least hundred days after the last study treatment administration. Female subjects who are breastfeeding should discontinue nursing prior to the first dose of study treatment and until at least hundred days after the last study treatment administration.

Exclusion Criteria:

* Use of any investigational agents ≤ 4 weeks before the planned day of leukapheresis.
* Concomitant malignancy or history of another malignancy (unless the Investigator rationalizes otherwise)
* Known concomitant presence of any active immunosuppressive disease (e.g. HIV) or any active autoimmune condition, except for vitiligo
* Any pre-existing contra-indication for contrast-enhanced MRI
* Pregnant or breastfeeding
* Any other condition, either physical or psychological, or reasonable suspicion thereof on clinical or special investigation, which contraindicates the use of the vaccine, or may negatively affect patient compliance, or may place the patient at higher risk of potential treatment complications

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of leukapheresis in pediatric patients with HGG and DIPG | Vaccine production and quality testing (i.e. from leukapheresis until 4 weeks after)
  Proportion of patients in the intention-to-treat (ITT) population that had successful leukapheresis
Feasibility of WT1-targeted DC vaccine production | Vaccine production and quality testing (i.e. from leukapheresis until 4 weeks after)
  Proportion of patients in the ITT population that had successful vaccine production (i.e. production of 9 or more vaccine doses meeting quality control requirements)
Feasibility of DC vaccine administration in pediatric patients with HGG and DIPG (administration of 1st vaccine) | At the administration of the 1st vaccine (i.e. +- 2 months after leukapheresis)
  Proportion of efficacy evaluable patients (i.e. having received at least 1 vaccine + no major protocol violation) in the intention-to-treat (ITT) population
Feasibility of DC vaccine administration in pediatric patients with HGG and DIPG according to the study treatment schedule | Study treatment scheme (i.e. from leukapheresis to administration of the 9th vaccine, +- 34 weeks)
  Proportion of patients in the ITT population who completed the study treatment (i.e. from leukapheresis until administration of the 9th vaccine)
Safety of DC vaccine administration in pediatric patients with HGG and DIPG: Related (Severe) Adverse Events ((S)AEs) | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later)
  Proportion of patients of the safety population that experienced (S)AEs possibly, probably or definitely related to DC vaccination
Safety of DC vaccine administration in pediatric patients with HGG and DIPG: total (S)AEs (number) | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later)
  Number of (S)AEs in the safety population (i.e. having received at least 1 DC vaccine)
Safety of DC vaccine administration in pediatric patients with HGG and DIPG: total (S)AEs (grade) | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later)
  Grade of (S)AEs in the safety population

SECONDARY OUTCOMES:
Indicators of clinical efficacy: Best overall response (BOR) | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later).
  BOR will be determined per patient as the best response designation over the study, based on radiologic RANO criteria. The response categories are: complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD).
Indicators of clinical efficacy: Progression-free survival (PFS) | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later). PFS may be updated after study completion.
  PFS is defined as the time (in months) between diagnosis/study entry and the date of progression (recurrence in the case of total resection) or death due to any cause, whichever occurs first.
Indicators of clinical efficacy: Overall survival (OS) | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later). OS may be updated after study completion.
  OS is defined as the time (in months) between diagnosis/study entry and death due to any cause.
Immunogenicity of vaccination with WT1-targeted DC in pediatric patients with HGG and DIPG: occurrence of WT1-specfic CD8+ T cells | On the day of the 1st (about 2 months after leukapheresis), 4th (about 3 months after leukapheresis) and 7th DC vaccine (about 6 months after leukapheresis)
  Occurrence of WT1-specific CD8+ T cells as assessed by tetramer staining (% positive cells)
Immunogenicity of vaccination with WT1-targeted DC in pediatric patients with HGG and DIPG: occurrence of WT1-specfic CD8+ T cells | On the day of the 1st (about 2 months after leukapheresis), 4th (about 3 months after leukapheresis) and 7th DC vaccine (about 6 months after leukapheresis)
  Occurrence of WT1-specific CD8+ T cells as assessed by TCR sequencing
Immunogenicity of vaccination with WT1-targeted DC in pediatric patients with HGG and DIPG: Functional WT1-specific T cell responses | On the day of the 1st (about 2 months after leukapheresis), 4th (about 3 months after leukapheresis) and 7th DC vaccine (about 6 months after leukapheresis)
  Functional WT1-specific T cell responses as assessed by multiparametric flow cytometry following antigen-specific stimulation (% positive cells)
Evaluation of changes in quality of life: How patients experience different phases of the study treatment schedule | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later)
  PedsQL Generic core scale and PedsQL Cancer Module. Higher scores indicate better health-related quality of life/lower problems.
Evaluation of changes in quality of life: How patient- and proxy-reported disease-related symptoms evolve over time during the study | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later)
  PedsQL Cancer Module. Higher scores indicate lower problems.
Evaluation of changes in quality of life: How patient- and proxy-reported general quality of life evolves over time during the study | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later)
  PedsQL Generic core scale. Higher scores indicate better health-related quality of life.

OTHER OUTCOMES:
Biomarker identification | over the entire study duration (i.e. from inclusion to end of follow-up, which lasts until 90 days after the last DC vaccine, or 24 months after inclusion, whichever occurs later)
  By means of associative analyses with clinical response and outcome, biomarkers will be identified among immunological parameters and tumor characteristics (if homogeneity of population allows).
Evaluation of changes in executive function | at baseline, upon completion of the study treatment scheme (i.e. after the 9th DC vaccine), at progression (if applicable) and 90 days after the final DC vaccine
  By means of BRIEF (Behavior Rating Inventory of Executive Function) questionnaires, completed before and after the study treatment scheme, it will be assessed how the patient's executive function changes from baseline. Higher T scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zwi N Berneman, MD, PhD, Principal Investigator — Antwerp University Hospital, Division of Hematology and Center for Cell Therapy and Regenerative Medicine
Locations (1):
- Unitversity Hospital Antwerp, Edegem, Belgium

REFERENCES:
- [Background] Van Tendeloo VF, Ponsaerts P, Lardon F, Nijs G, Lenjou M, Van Broeckhoven C, Van Bockstaele DR, Berneman ZN. Highly efficient gene delivery by mRNA electroporation in human hematopoietic cells: superiority to lipofection and passive pulsing of mRNA and to electroporation of plasmid cDNA for tumor antigen loading of dendritic cells. Blood. 2001 Jul 1;98(1):49-56. doi: 10.1182/blood.v98.1.49. PMID 11418462
- [Background] Van Tendeloo VF, Van de Velde A, Van Driessche A, Cools N, Anguille S, Ladell K, Gostick E, Vermeulen K, Pieters K, Nijs G, Stein B, Smits EL, Schroyens WA, Gadisseur AP, Vrelust I, Jorens PG, Goossens H, de Vries IJ, Price DA, Oji Y, Oka Y, Sugiyama H, Berneman ZN. Induction of complete and molecular remissions in acute myeloid leukemia by Wilms' tumor 1 antigen-targeted dendritic cell vaccination. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13824-9. doi: 10.1073/pnas.1008051107. Epub 2010 Jul 14. PMID 20631300
- [Background] Benteyn D, Anguille S, Van Lint S, Heirman C, Van Nuffel AM, Corthals J, Ochsenreither S, Waelput W, Van Beneden K, Breckpot K, Van Tendeloo V, Thielemans K, Bonehill A. Design of an Optimized Wilms' Tumor 1 (WT1) mRNA Construct for Enhanced WT1 Expression and Improved Immunogenicity In Vitro and In Vivo. Mol Ther Nucleic Acids. 2013 Nov 19;2(11):e134. doi: 10.1038/mtna.2013.54. PMID 24253259
- [Background] Van Driessche A, Berneman ZN, Van Tendeloo VF. Active specific immunotherapy targeting the Wilms' tumor protein 1 (WT1) for patients with hematological malignancies and solid tumors: lessons from early clinical trials. Oncologist. 2012;17(2):250-9. doi: 10.1634/theoncologist.2011-0240. Epub 2012 Jan 30. PMID 22291091
- [Background] Anguille S, Smits EL, Bryant C, Van Acker HH, Goossens H, Lion E, Fromm PD, Hart DN, Van Tendeloo VF, Berneman ZN. Dendritic Cells as Pharmacological Tools for Cancer Immunotherapy. Pharmacol Rev. 2015 Oct;67(4):731-53. doi: 10.1124/pr.114.009456. PMID 26240218
- [Background] Anguille S, Van de Velde AL, Smits EL, Van Tendeloo VF, Juliusson G, Cools N, Nijs G, Stein B, Lion E, Van Driessche A, Vandenbosch I, Verlinden A, Gadisseur AP, Schroyens WA, Muylle L, Vermeulen K, Maes MB, Deiteren K, Malfait R, Gostick E, Lammens M, Couttenye MM, Jorens P, Goossens H, Price DA, Ladell K, Oka Y, Fujiki F, Oji Y, Sugiyama H, Berneman ZN. Dendritic cell vaccination as postremission treatment to prevent or delay relapse in acute myeloid leukemia. Blood. 2017 Oct 12;130(15):1713-1721. doi: 10.1182/blood-2017-04-780155. Epub 2017 Aug 22. PMID 28830889
- [Background] Z. Berneman, A. Van de Velde, S. Anguille, Y. Willemen, M. Huizing, P. Germonpré, K. Saevels, G. Nijs, N. Cools, A. Van Driessche, B. Stein, H. De Reu, W. Schroyens, A. Gadisseur, A. Verlinden, K. Vermeulen, M. Maes, M. Lammens, H. Goossens, M. Peeters, V. Van Tendeloo, E. Smits. Vaccination with Wilms' Tumor Antigen (WT1) mRNA-Electroporated Dendritic Cells as an Adjuvant Treatment in 60 Cancer Patients: Report of Clinical Effects and Increased Survival in Acute Myeloid Leukemia, Metastatic Breast Cancer, Glioblastoma and Mesothelioma. Cytotherapy 2016, 18(6), p. S13-14
- [Background] Z. Berneman, S. Anguille, Y. Willemen, A. Van de Velde, P. Germonpré, M. Huizing, V. Van Tendeloo, K. Saevels, L. Rutsaert, K. Vermeulen, A. Snoeckx, B. Op de Beeck, N. Cools, G. Nijs, B. Stein, E. Lion, A. van Driessche, M. Peeters, E. Smits. Vaccination of cancer patients with dendritic cells electroporated with mRNA encoding the Wilms' Tumor protein (WT1): correlation of clinical effect and overall survival with T-cell response. Cytotherapy 2019, 21(5), p. S10.
- [Background] de Bruijn S, Anguille S, Verlooy J, Smits EL, van Tendeloo VF, de Laere M, Norga K, Berneman ZN, Lion E. Dendritic Cell-Based and Other Vaccination Strategies for Pediatric Cancer. Cancers (Basel). 2019 Sep 19;11(9):1396. doi: 10.3390/cancers11091396. PMID 31546858
- [Background] Benitez-Ribas D, Cabezon R, Florez-Grau G, Molero MC, Puerta P, Guillen A, Paco S, Carcaboso AM, Santa-Maria Lopez V, Cruz O, de Torres C, Salvador N, Juan M, Mora J, La Madrid AM. Immune Response Generated With the Administration of Autologous Dendritic Cells Pulsed With an Allogenic Tumoral Cell-Lines Lysate in Patients With Newly Diagnosed Diffuse Intrinsic Pontine Glioma. Front Oncol. 2018 Apr 26;8:127. doi: 10.3389/fonc.2018.00127. eCollection 2018. PMID 29755954
- [Background] Lasky JL 3rd, Panosyan EH, Plant A, Davidson T, Yong WH, Prins RM, Liau LM, Moore TB. Autologous tumor lysate-pulsed dendritic cell immunotherapy for pediatric patients with newly diagnosed or recurrent high-grade gliomas. Anticancer Res. 2013 May;33(5):2047-56. PMID 23645755
- [Derived] Van Genechten T, De Laere M, Van den Bossche J, Stein B, De Rycke K, Deschepper C, Hazes K, Peeters R, Couttenye MM, Van De Walle K, Roelant E, Maes S, Vanden Bossche S, Dekeyzer S, Huizing M, Caluwaert K, Nijs G, Cools N, Verlooy J, Norga K, Verhulst S, Anguille S, Berneman Z, Lion E. Adjuvant Wilms' tumour 1-specific dendritic cell immunotherapy complementing conventional therapy for paediatric patients with high-grade glioma and diffuse intrinsic pontine glioma: protocol of a monocentric phase I/II clinical trial in Belgium. BMJ Open. 2024 Mar 18;14(3):e077613. doi: 10.1136/bmjopen-2023-077613. PMID 38503417
- See also: Related Info — https://www.uza.be/CCRG